CLINICAL TRIAL: NCT03631550
Title: The RIME Study - Combined Occipital and Supraorbital Transcutaneous Nerve Stimulation for Treatment of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurolief Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-302 RIME
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Acute Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): Relivion Active device
  Interventions: Device: Relivion active
- Sham (Sham Comparator): Relivion Sham device
  Interventions: Device: Relivion Sham

INTERVENTIONS:
Device: Relivion active — 1 hour self-administered occipital and supraorbital transcutaneous nerve stimulation
  Arms: Active
Device: Relivion Sham — 1 hour self-administered Sham occipital and supraorbital transcutaneous nerve stimulation
  Arms: Sham

SUMMARY:
this study will evaluate the clinical performance and safety of a self administered abortive treatment for migraine headache using combined occipital and supraorbital transcutaneous nerve stimulator (Neurolief device, Relivion®)

DETAILED DESCRIPTION:
The Relivion® is a non-invasive transcutaneous neuro-stimulator is indicated for the acute treatment of migraine with or without aura in subjects 18 years of age or older. The Relivion® is intended to be a prescription device, self-used at home.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age and older.
2. Subject meets the ICHD (International Classification of Headache Disorders)-3 (2018) diagnostic criteria for Migraine with or without aura.
3. Subject reports 1-6 Migraine attacks per month; other headaches no more than 6 days per month.
4. Subject is willing to and capable of complying with the specified study requirements, provided written Informed Consent, can complete the electronic diaries, and can be contacted by telephone.

Exclusion Criteria:

1. Subject having received Botox treatment in the head region in the prior 3 months.
2. Subject having received supraorbital or occipital nerve blocks in the prior month.
3. Past 6 months of chronic migraine, New Daily Persistent Headache, and chronic tension-type headache per ICHD-3 (2018) diagnostic criteria.
4. Current medication overuse headache.
5. Use of opioid medications in the prior 1 month.
6. Use of barbiturates in the prior 1 month.
7. Subject has >10 headache days per month
8. Implanted metal/shrapnel or electrical devices in the head (not including dental implants), a cardiac pacemaker or an implanted or wearable defibrillator.
9. Received parenteral infusions for migraine within the previous 2 weeks.
10. Subject has known uncontrolled epilepsy.
11. History of neurosurgical interventions
12. Subject with implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
13. Current drug abuse or alcoholism.
14. Subject is participating in any other clinical study.
15. Skin lesion or inflammation at the region of the stimulating electrodes.
16. Personality or somatoform disorder.
17. Pregnancy or Lactation.
18. Women with child bearing potential without medically acceptable method of contraception (NOTE: Females of child bearing potential must have a negative pregnancy test).
19. Documented history of cerebrovascular event.
20. Subject with recent brain or facial trauma (occurred less than 3 months prior to this study).
21. Subject participated in a previous study with the Relivion device.
22. The subject does not have the basic cognitive and motor skills needed to operate a smartphone.
23. Subject with head circumference smaller than 51 centimeters or head circumference larger than 60 centimeters
24. Subject with other significant pain problem that in the opinion of the investigator may confound the study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: stewart J. Tepper, Dr., Principal Investigator — Dartmouth-Hitchcock Medical Center, Lebanon, NH, USA
Locations (12):
- United States (6):
  - Clinical Research Consortium, an AMR company, Tempe, Arizona
  - Hartford HealthCare Headache Center, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Regeneris Medical, North Attleboro, Massachusetts
  - Clinical Research Consortium, an AMR company, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
- Israel (6):
  - Barzilai MC, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Sharei Zedek MC, Jerusalem
  - Macabi healtcenter services, Kfar Saba
  - Laniado MC, Netanya
  - Macabi healtcenter services, Raanana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tepper SJ, Grosberg B, Daniel O, Kuruvilla DE, Vainstein G, Deutsch L, Sharon R. Migraine treatment with external concurrent occipital and trigeminal neurostimulation-A randomized controlled trial. Headache. 2022 Sep;62(8):989-1001. doi: 10.1111/head.14350. Epub 2022 Jun 24. PMID 35748757

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Sham
Started (Full Analysis set (FA) include all the subjects randomized, including the subjects treated with the device up to May 31, 2019) | 94 | 93
The ITT Analysis Set (The Intent to Treat (ITT) analysis set which includes all randomized subjects who were treated with the device after May 31, 2019 (including self-practice). Per ITT principles, all subjects were analyzed as randomized.) | 67 | 64
The mITT Analysis Set (The mITT analysis set which includes all subjects from the ITT analysis set who treat at least one eligible attack (excluding the "self-practice test") analyzed as treated.) | 50 | 59
Completed (from FA set) | 67 | 64
Not Completed | 27 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 64 | 130
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (12.47) | 39.9 (13.03) | 40.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 51 | 109
  Male | 9 | 13 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 60 | 57 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 24 | 53
  Israel | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Reporting Reduction of Migraine Headache Pain at 2 Hours From Treatment Initiation
Description: the number and percent of subjects reporting reduction of migraine headache pain 2 hours post treatment initiation from severe or moderate to mild or no pain, or from mild to no pain, in their first eligible treated migraine attack (if rescue therapy was not used)
Time Frame: 2 hours from treatment initiation
Population: mITT present the number and percentage of subjects with pain relief (reduction in pain level) 2 hours post-treatment, from severe or moderate to mild or no pain, or from mild to no pain, in their first eligible treated episode. If a subject had used rescue medication up to the assessment time point, he/she was considered as not reaching the endpoint. mITT set included 50 patients in the Active arm and 59 patients in the sham arm
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 50 | 59
Participants | 30 | 22
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p = 0.018, Chi-squared

2. Secondary Outcome: Proportion of Subjects Reporting Improvement in Their Most Bothersome Symptom (MBS) Other Than a Headache, 2 Hours Post-treatment Initiation
Description: The number and percentage of subjects reporting improvement in their Most Bothersome Symptom (MBS) other than a headache, 2 hours post-treatment initiation (if rescue therapy was not used), in their first eligible treated migraine attack. MBS may be nausea, photophobia, phonophobia
Time Frame: 2 hours from treatment initiation
Population: mITT population analysis. mITT set included 50 patients in the Active arm from which 36 reported MBS and 59 patients in the sham arm from which 45 reported MBS
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 36 | 45
Participants | 29 | 27
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p = 0.0466, Chi-squared

3. Secondary Outcome: Proportion of Subjects Reporting Reduction of Migraine Headache Pain 1-hour Post Treatment Initiation
Description: The number and percentage of subjects reporting reduction of migraine headache pain 1-hour post treatment initiation (if rescue therapy was not used), from severe or moderate to mild or no pain, or from mild to no pain, in their first eligible treated migraine attack
Time Frame: 1 hour from treatment initiation
Population: mITT population analysis. mITT set included 50 patients in the Active arm and 59 patients in the sham arm
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 50 | 59
Participants | 21 | 15
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p = 0.0677, Chi-squared

4. Secondary Outcome: Proportion of Subjects Who Are Pain Free at 2 Hours Post Treatment Initiation
Description: The number and percentage of subjects who are pain free at 2 hours post treatment initiation (if rescue therapy was not used), in their first eligible treated migraine attack
Time Frame: 2 hours from treatment initiation
Population: mITT population anaylsis. mITT set included 50 patients in the Active arm and 59 patients in the sham arm
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 50 | 59
Participants | 23 | 7
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p < .0001, Chi-squared

5. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Safety of the study device following study treatment: Number and Rate of participates with Adverse events related or unrelated to the study device
Time Frame: From Enrollment (randomization) through study exit i.e. 70 days
Population: ITT population analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 67 | 64
Participants
  Participants with Adverse Events | 8 | 2
  Participants with device related Adverse Events | 5 | 2
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Other; p = 0.0968, Fisher Exact

6. Other Pre Specified Outcome: The Change in Pseudo-continuous Pain Score From Baseline to 1-hour Post Treatment
Description: as per the Statistical Considerations for Clinical Trials During the COVID-19 Public Health Emergency" June 2020 FDA Guidance, which states that a modifications to the definition and ascertainment of trial endpoints may be warranted to address the impact of COVID-19. A potential modification for a binary endpoint that is based on a continuous or ordinal measurement is by using the continuous or ordinal measurement as the endpoint. therefore, an additional analysis to the study end points , the migraine headache pain level was transformed into a numerical score (pseudo-continuous): "No pain"=0, "Mild"=1, "Moderate"=2, "Severe"=3. If rescue medication was used, the score after the rescue intake post-treatment are set to the baseline value. The change from baseline is compared between the study arms with an analysis of covariance model adjusted for site and baseline pain level.
Time Frame: baseline to 1-hour post treatment
Population: mITT set included 50 patients in the Active arm and 59 patients in the sham arm
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 50 | 59
units on a scale | -0.637 [-0.881 to -0.392] | -0.306 [-0.537 to -0.075]
Statistical Analysis 1: Comparison: Active vs Sham; Test type: Superiority; p = 0.0121, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events data were collected per study participant from Enrollment (randomization) through study exit. ie 70 days
Description: Adverse events related or unrelated to the study device and/or procedure were collected per study participant from Enrollment (randomization) through study exit. The ITT data analysis set served as the principal data analysis set for the safety analyses.
Arm/Group | Active | Sham
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/64
Other Adverse Events (participants affected / at risk) | 8/67 | 2/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=67) | Sham (N=64)
Migraine (Nervous system disorders) | 1 (2) | 0 (0)
Unpleasant sensation during treatment (Nervous system disorders) | 1 (1) | 1 (3)
Scalp numbness sensation (Nervous system disorders) | 1 (1) | 0 (0)
Pain (Nervous system disorders) | 1 (2) | 0 (0)
Skin redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Tingling (Nervous system disorders) | 1 (1) | 0 (0)
Twitching (Nervous system disorders) | 1 (1) | 0 (0)
COVID (Infections and infestations) | 1 (1) | 0 (0)
upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
inner ear scratch (Ear and labyrinth disorders) | 1 (1) | 0 (0)
lip numbness (General disorders) | 1 (1) | 0 (0)
Pressure/discomfort of head (Nervous system disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT03631550/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT03631550/SAP_001.pdf